CLINICAL TRIAL: NCT06710821
Title: Phase I Clinical Study of Irinotecan Liposomes in Combination with Temozolomide and Vincristine in the Treatment of Patients with Relapsed/refractory Pediatric Solid Tumors
Brief Title: Irinotecan Liposomes Combined with Temozolomide and Vincristine in the Treatment of Pediatric Patients with Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY- SARC-GD01
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor Cancer
Keywords: Adolescent; solid tumors; VIT
MeSH Terms: interventions — irinotecan sucrosofate; Vincristine; Temozolomide

STUDY DESIGN:
Intervention Model Description: Irinotecan liposome combined with temozolomide and vincristine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VIT (Experimental): Vincristine: 1.5 mg/m², iv, d1. l Temozolomide 150 mg/m²/d, iv drip, d1-5. l Irinotecan liposomal RP dose, iv infusion over 90 min, d1.
  Interventions: Drug: Liposomal irinotecan in combination with vincristine and temozolomide

INTERVENTIONS:
Drug: Liposomal irinotecan in combination with vincristine and temozolomide — Vincristine: 1.5 mg/m², iv, d1. l Temozolomide 150 mg/m²/d, iv drip, d1-5. l Irinotecan liposomal RP dose, iv infusion over 90 min, d1. Q3W, 4 cycles expected until disease progression or intolerable toxicity occurs

SUMMARY:
A prospective, single-center Ia/Ib clinical study divided into two parts, including Phase Ia Dose Exploration and Phase Phase Ib Extension Phase.

DETAILED DESCRIPTION:
Phase Ia dose exploration phase:

Using a "3+3" study design, 15-30 eligible subjects will receive irinotecan liposome. Five dose groups of irinotecan liposome 40 mg/m2, 50 mg/m2, 65 mg/m2, 80 mg/m2, and 100 mg/m2 will be pre-determined for a 21-day cycle. The dose of liposomal irinotecan will be gradually increased from the low dose group to the high dose group, and DLT will be observed during the dosing cycle.The same subject will receive only one dose of liposomal irinotecan during the study period. All subjects will complete relevant protocol-specified investigations during the course of treatment to observe safety and initial efficacy.

Phase Ib Expansion Phase:

Based on the results of the Phase Ia dose-climbing phase, the Phase Ib study will be conducted at the RP dose of irinotecan liposomes, and all subjects will complete the relevant examinations specified in the protocol during treatment to observe safety, preliminary efficacy, and so on.

ELIGIBILITY:
Inclusion Criteria:

* 1、 12 years old ≤ 18 years old, no gender restriction.
* 2. Karnofsky (≥ 16 years old) or Lansky (< 16 years old) physical condition score of at least 50.
* 3. Expected survival time of at least 12 weeks.
* 4.Cardiac function: A) LVEF ≥50% by cardiac ultrasound; B) no myocardial ischemia by electrocardiogram; C) no history of arrhythmia requiring pharmacological intervention before enrollment.
* 5、 Patients who met the clinical diagnostic criteria and were diagnosed with solid malignant tumors in children; and 6, Patients who have progressed, relapsed, or are refractory to first-line therapy (failed to achieve complete or partial remission after recent treatment); and
* 7, Measurable lesions (according to RECIST 1.1 criteria, CT/MRI scan length of tumor lesions ≥ 10mm, CT/MRI scan short diameter of lymph node lesions ≥ 15mm, measurable lesions have not received local treatment such as radiotherapy, cryotherapy, etc.); patients with neuroblastoma, at least one of which is diagnosed by Computed Tomography (CT), Magnetic Resonance Imaging (MRI), and/or by Bone Marrow ( BM) morphology and/or a measurable lesion by mesoiodobenzylguanidine (MIBG) scan obtained within 4 weeks of enrollment (MRI or CT scan or X-ray measurable tumor);
* 8. Patients must have fully recovered from the acute toxic effects of all prior anticancer chemotherapy: A) Myelosuppressive chemotherapy: at least 21 days (42 days if nitrosourea was used previously) after the last myelosuppressive chemotherapy, including cytotoxic drugs given in a low-dose rhythmic regimen; B) Experimental drugs or anticancer treatments other than chemotherapy: not available for 28 days prior to the planned start of AI or VIT Use. Complete recovery from clinically significant toxicity of the treatment must be established; C) Hematopoietic Growth Factors: at least 14 days after the last administration of long-acting growth factors or 3 days after the last administration of short-acting growth factors; D) Immunotherapies: at least 42 days after completion of any type of immunotherapy (other than steroids), such as immune checkpoint inhibitors and tumor vaccines; E) X-Ray Therapy (XRT): local palliative E) X-Ray Therapy (XRT): at least 14 days after localized palliative XRT (small-bore); for other substantial bone marrow (BM) irradiation, must be completed at least 42 days; F) Stem Cell Infusion without Total Body Irradiation (TBI): no evidence of active graft-versus-host disease, and the transplantation or stem cell infusion must be completed at least 56 days after the infusion.
* 9. Laboratory tests at screening should fulfill the following conditions: A) Absolute neutrophil (ANC) ≥1.5×109/L (ANC ≥1.0×109/L if bone marrow infiltration); B) Platelet count (PLT) ≥75×109/L (bone marrow infiltration PLT ≥50×109/L); C) Bilirubin (combined + uncombined total) ≤1.5 upper limit of normal ( ULN), and patients with confirmed diagnosis of Gilbert's syndrome may be included in this group at the investigator's discretion; D) estimated glomerular filtration rate ≥30 mL/min/1.73 m2 or serum creatinine (Cr) ≤1.5 ULN (calculated according to the standard Cockcroft-Gault formula); E) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (5 times the ULN if liver metastases are present)
* 10. be able to comply with outpatient treatment, laboratory monitoring, and required clinical visits during the study period; and
* 11. Parents/guardians of child or adolescent subjects are able to understand, agree to, and sign the study Informed Consent Form (ICF) and applicable Child Consent Form prior to initiation of any program-related procedures; subjects are able to give consent with parental/guardian consent (if applicable).

Exclusion Criteria:

* 1, Patients who have received prior irinotecan in combination with temozolomide and vincristine, or who have progressed after receiving irinotecan or temozolomide; and
* 2, P450 enzyme-inducing anticonvulsants (anticonvulsants affect irinotecan clearance); and
* 3. Active cardiovascular disease of previous or concurrent clinical significance, including congenital heart disease or pericardial disease, history of heart failure, myocardial infarction, coronary artery disease, cardiac valve disease, cardiomyopathy, cardiac arrhythmias (including persistent atrial fibrillation, complete left bundle-branch block, and frequent premature ventricular episodes); or prolongation of the QT interval (QTc)> after the current corrected heart rate of 480 milliseconds; and cardiac function classified according to the New York Heart Association (NYHA). NYHA cardiac function classification (age > 3 years) or infant cardiac function criteria (age ≤ 3 years) or class III-IV cardiac insufficiency with a left ventricular ejection fraction (LVEF) < 50%, as indicated by color Doppler echocardiography; and
* 4. Prior severe chronic skin disease; and
* 5, Previous allergic asthma or severe allergic disease; 6, Uncontrolled hypertension and diabetes mellitus; and
* 6. Poorly controlled hypertension and diabetes mellitus.
* 7. History of other tumors, except cervical cancer or basal cell carcinoma of the skin that has been cured; 8.
* 8. Hepatitis B surface antigen positive patients; and
* 9. Patients with HIV or syphilis infection; and
* 10. Patients who have previously received an organ transplant; and
* 11. Uncontrolled and active systemic bacterial, viral or fungal infections.
* 12. Contraindications to the use of high-dose hormones, such as uncontrolled hyperglycemia, gastric ulcers, or psychiatric disorders; and
* 13. History of severe neurologic or psychiatric disorders, including epilepsy or autism;
* 14. Patients who, in the judgment of the investigator, are not suitable for participation in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 6 months
  maximum tolerated dose (MTD) of liposomal irinotecan in combination with temozolomide and vincristine in pediatric patients with relapsed/refractory pediatric solid tumors

SECONDARY OUTCOMES:
Incidence of adverse events | 1 year
  Use NCI-CTCAE version 5.0 for classification and grading
Objective Response Rate | 1 year
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1

IPD SHARING:
Plan to Share IPD: No